CLINICAL TRIAL: NCT01719432
Title: Effect of Body Mass on Filgrastim Pharmacokinetics
Status: Completed | Type: Observational
Sponsor: Aaron Cumpston, PharmD, BCOP (Other)
Responsible Party: Sponsor-Investigator, Aaron Cumpston, PharmD, BCOP, Clinical Specialist - BMT, West Virginia University
Organization: West Virginia University (Other)
Other Study IDs: WVU 021112
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hematological Malignancy; Neutropenia
Keywords: Filgrastim; Obese; Non-obese; Pharmacokinetics
MeSH Terms: conditions — Hematologic Neoplasms; Neutropenia; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obese patients
- Non-obese patients

SUMMARY:
Studies have shown that different percentages of body fat can alter the way drugs are distributed in the body. This study will use blood samples taken at different time points for patients taking Neupogen to determine if higher body weights affect drug exposure. The information gathered from this study will help understand if patients with higher body weights need a different dosing plan.

Patients in this study will have blood draws once before they take Neupogen and 6 times after they take the Neuopen (for a total of 24 hours). These patients will be in the hospital already and will not need to make additional trips back to have blood drawn. A total of about 5-6 tablespoons of blood will be drawn for this study. 15 obese patients and 15 matched, non-obese patients will be enrolled into this study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Receiving filgrastim at 5mcg/kg ± 10%
* Admitted as an inpatient with an expected stay of at least 24 hours
* Weight is > 190% of their ideal body weight (IBW) for "obese" patients or within 80 - 124% of IBW for matched control patients.
* Patient or their legally authorized representative understands and voluntarily signs the written informed consent prior to any study-specific procedures. A copy of the signed informed consent form will be retained by the treating institution.

Exclusion Criteria:

* Patients who have received filgrastim within 24 hours prior to enrollment
* Patients who have received pegfilgrastim within 14 days prior to enrollment
* Hypersensitivity reaction to filgrastim or any related product
* Patients who have taken lithium within 7 days of enrollment
* Serum Creatinine > 1.5 mg/dL
* Patients who are pregnant or breastfeeding
* Patients who are unable to understand and/or render informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese and non-obese patients receiving filgrastim
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Systemic clearance of filgrastim in obese and non-obese patients | 24 hours

SECONDARY OUTCOMES:
Alpha and beta half-life of filgrastim in obese and non-obese patients | 24 hours
Maximum concentration (Cmax) of filgrastim in obese and non-obese patients | 24 hours
Time to maximum concentration (Tmax) of filgrastim in obese and non-obese patients | 24 hours
Volume of distribution (Vds and Vdss)of filgrastim in obese and non-obese patients | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Cumpston, PharmD, BCOP, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

REFERENCES:
- [Derived] Stewart AW, Shillingburg A, Petros W, Wen S, Piktel D, Moses R, Gibson LF, Craig M, Cumpston A. A prospective study of filgrastim pharmacokinetics in morbidly obese patients compared with non-obese controls. Pharmacotherapy. 2022 Jan;42(1):53-57. doi: 10.1002/phar.2646. Epub 2021 Nov 22. PMID 34767652